CLINICAL TRIAL: NCT04007263
Title: A Phase 1, Randomized, Double Blind, Multiple Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of NP10679 in Healthy Adults"
Brief Title: A Multiple Ascending Dose Study of Safety and Pharmacokinetics of NP10679 in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurop Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Pharmaron (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP10679-002; 3R44NS071657-06 (NIH)
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-07

CONDITIONS: Stroke, Ischemic; Pain, Postoperative; Substance Abuse; Subarachnoid Hemorrhage
Keywords: NMDA; GluN2B
MeSH Terms: conditions — Ischemic Stroke; Pain, Postoperative; Substance-Related Disorders; Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo intravenous infusion over 30 minutes, five days of once daily dosing
  Interventions: Drug: Placebo
- NP10679 25 mg (Experimental): NP10679 25 mg intravenous infusion over 30 minutes, five days of once daily dosing
  Interventions: Drug: NP10679
- NP10679 50 mg (Experimental): NP10679 50 mg intravenous infusion over 30 minutes, five days of once daily dosing
  Interventions: Drug: NP10679
- NP10679 100 mg (Experimental): NP10679 100 mg intravenous infusion over 30 minutes, five days of once daily dosing
  Interventions: Drug: NP10679

INTERVENTIONS:
Drug: Placebo — Placebo via 30 minute infusion once daily for 5 days
  Arms: Placebo
Drug: NP10679 — NP10679 25 mg via 30 minute infusion once daily for 5 days
  Arms: NP10679 100 mg; NP10679 25 mg; NP10679 50 mg

SUMMARY:
This multiple ascending dose study assesses the safety, tolerability and pharmacokinetics of NP10679 when delivered intravenously in escalating dose levels in comparison to placebo.

DETAILED DESCRIPTION:
NP10679 is a pH dependent inhibitor of the GluN2B subtype of the NMDA receptor. Compounds of this drug class are hypothesized to be beneficial in a number of central nervous system disorders, including brain ischemia associated with stroke, subarachnoid hemorrhage, severe pain, major depression and substance abuse disorders. This study uses a double blind, adaptive design approach to evaluate the safety, tolerability and pharmacokinetics of 5 once daily doses of NP10679 when delivered intravenously in three escalating dose levels in comparison to placebo

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 55 years
* Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.
* If of child bearing potential (both men and women) must agree to use 2 forms of contraceptive methods for the duration of study.

Exclusion Criteria:

* Clinical laboratory values greater than or equal to 2 times the upper limit of normal.
* Recent history (within 2 yrs) or current tobacco use.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events as a measure of safety and tolerability | 10 days
  Observed side effects and alteration in laboratory values
Plasma concentration of parent drug | 9 days
  Pharmacokinetic parameters during dosing period through 4 days post dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zaczek R, Traynelis SF, Dingledine R, Koszalka GW, Laskowitz DT. Phase 1 Clinical Results for NP10679, a pH-sensitive GluN2B-selective N-methyl-d-aspartate Receptor Inhibitor. Clin Pharmacol Drug Dev. 2023 Jul;12(7):706-717. doi: 10.1002/cpdd.1217. Epub 2023 Jan 15. PMID 36642931